CLINICAL TRIAL: NCT07274189
Title: Maintenance of Periodontal Health With Daily Use of Sodium Bicarbonate Toothpaste
Brief Title: Periodontal Health and Sodium Bicarbonate Toothpaste
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Collaborators: HALEON (Industry)
Responsible Party: Principal Investigator, Zoe Brookes, Associate Head of School (Teaching & Learning), University of Plymouth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5350
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-09

CONDITIONS: Periodontal Diseases
Keywords: periodontitis; periodontal disease; sodium bicarbonate; toothpaste; microbiome
MeSH Terms: conditions — Periodontal Diseases; Periodontitis | interventions — BaseLine dental cement

STUDY DESIGN:
Intervention Model Description: N/A, care pathway follows national guidelines.
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium bicarbonate toothpaste (67%) (Active Comparator): Description: Intervention includes receiving Corsodyl Complete Protection Extra Fresh Toothpaste to use which contains sodium bicarbonate.
  Interventions: Procedure: no treatment received; Procedure: Periodontal treatment and OHI
- Fluoride toothpaste (1450ppm) (Sham Comparator): Control group to receive Aquafresh Fresh and Minty Toothpaste
  Interventions: Procedure: no treatment received; Procedure: Periodontal treatment and OHI

INTERVENTIONS:
Procedure: no treatment received — Baseline; 0 months (no periodontal treatment)
  Other Names: Gum treatment (baseline)
Procedure: Periodontal treatment and OHI — 3 months periodontal treatment & OHI
  Other Names: Gum treatment (3 mons)
Procedure: Periodontal treatment and OHI — 6 months periodontal treatment & OHI
  Other Names: Gum treatment (6 mons)

SUMMARY:
The goal of this clinical trial is to determine whether sodium bicarbonate fluoride toothpaste can help maintain periodontal health in adults who have undergone non-surgical periodontal treatment. The main question it aims to answer is:

Does daily use of toothpaste affect the following outcomes: clinical oral health (plaque scores, gingival bleeding scores and periodontal pocket depths), salivary biochemical markers and the oral microbiome.

Outcomes measures will be recorded at 0,3, and 6 months, during which time participants will receive either the treatment or placebo toothpaste and undergo oral hygiene instruction and PMPR over 6 months.

DETAILED DESCRIPTION:
Study Design, Setting and Participants

The investigators will conduct an ongoing longitudinal study evaluating structured hygiene treatment, with required dental treatment over six months, with outcome measures recorded at three time points: baseline (0 months), 3 months, and 6 months.

The study will recruit adult male and female individuals (n=100, aged >18 years) from patients attending Peninsula Dental School (PDS) Dental Education Facilities in Plymouth.

These patients will not currently be being seen by students and therefore will be recruited to take part in a 6-month study, where their oral hygiene, periodontal treatment and dental treatment will be carried out by our research team.

Before completing recruitment and booking in for any dental appointments, the following exclusion criteria will applied to the patients: previous diagnosis of diabetes (Type I or II), current antibiotics use, complete denture users, immunosuppressants use, antimicrobial mouthwash use within 3 months.

Later exclusion criteria will be applied to patients after seeing the dentist, if they have a BPE score including less than one code 3 and/or more than two code 4's. The study is ongoing and is scheduled to conclude data collection in October 2026 at the latest.

Intervention The intervention will consist of one initial dental examination, three confirmed visits with the hygienist, and an additional unlimited number of dental appointments depending on the level of treatment each patient required within the 6-month research period the patient was on the trial.

Participants will receive standardised professional hygiene treatment consisting of sub- and supra-gingival Professional Mechanical Plaque Removal (PMPR), delivered by qualified hygienists.

Integrated dental care, including preventive and restorative interventions, will be provided as clinically indicated. Study visits are separate from student treatment schedules, ensuring no crossover of care outside the study protocol.

The study workflow involves.

* Initial Dental Appointment (30 minutes): Initial dental examination; visual oral inspection, BPE, radiographs (if required). Dental specific treatment plan created for each patient.
* Hygiene Appointment 1 (Baseline, 0 months): Written consent collected, along with a full medical and dental history. Blood pressure and saliva samples taken. Full periodontal assessment (FPA), plaques and bleeding scores measured. Oral Hygiene Instruction (OHI) and PMPR given. Oral hygiene home pack given to the patients including toothpaste and interdental brushes. The 3 month follow up appointment booked.
* Hygiene Appointment 2 (3 months): All measuerments repeated. OMS, BP, FPA, P, BOP, OHI review, PMPR. Oral hygiene home pack replenished. Next hygiene appointment booked for 3 months' time.
* Hygiene Appointment 3 (6 months;): All measurements completed. Patient discharged from research appointments.
* Additional Dental Treatment Appointments (as needed): The amount and duration of these dental treatment appointments varied depending on the individual needs of the patients within the study. However, these appointments generally will generally included extractions, restorations, dentures appointments, crowns and root canal treatments, i.e. anything the patients requires over the 6 months of the study, between hygiene appointments, to complete the course of treatment.

Clinical Workflow and Team Integration:

The study relies on coordinated interdisciplinary teamwork:

* Dental Hygienists: Deliver hygiene treatment, provide oral health counselling, and record clinical outcomes.
* Dentists: Oversee treatment, provide integrated dental care, and ensure patient safety.
* Dental Nurses: Support clinical procedures, maintain infection control, oral microbiome sample collection and manage documentation.
* Research Scientists: Overall project management, oversee protocol adherence, oral microbiome sample collection/analysis, and manage research data.
* Administrative Staff: Manage scheduling and patient communication.
* Expert Supervisors:

Data Collection and Outcomes:

Data will be collected and stored digitally for research purposes but also input into the patients R4 dental records. Paper copies of plaque and bleeding indices were also kept in paper format in the patients paper files along with copies of their consent.

Clinical data, including plaque index, gingival health, and periodontal parameters, will be recorded at each hygiene visit. Oral microbiome samples will be collected at all three hygiene time points to support parallel research objectives to quantify the following:

* Dental Parameters: Dental charting (DMFT), Basic Periodontal Examination (BPE), plaque and bleeding scores, and periodontal pocket/attachment measurements, with periodontitis severity classified using BSP guidelines.
* Oral Samples: Unstimulated saliva samples will be collected (unstimulated, 5 min) and stored at -80 °C. Saliva supernatant will be used for biochemical marker analysis (nitrate, nitrite, ammonia, pH, buffering capacity, lactate, glucose, interleukins), while salivary pellets will be used for oral microbiome analysis. Sodium nitrate (80 μmol) mouth rinse will be collected and stored at -80 °C. Mouth rise will be used quantification of oral nitrate reducing capacity.
* Blood Pressure (BP): blood pressure will be recorded from an average of 3 values following standard protocols. Participants BP results will be classified according to NICE and NHS guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants >18 years, of any gender will be recruited.

Exclusion Criteria:

* Full dentures
* Diabetics
* Cancer diagnosis
* Pregnancy
* Use of antibiotics (<3 months prior to participation)
* Use of antibacterial mouthwash
* Inorganic nitrates taken less than 4 weeks before the study
* Immunosuppressants taken less than 4 weeks before the study
* BPE's score of less than 3, and or/ BPE score of more than two 4's.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-10-20 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Maintenance of periodontal health | 6 months
  Determine whether sodium bicarbonate fluoride toothpaste as part of daily oral hygiene, can provide benefits for maintenance of clinical periodontal health post non-surgical periodontal treatment.

SECONDARY OUTCOMES:
Oral Microbiome Changes | 6 months
  Does the oral microbiome and biochemical composition of saliva differ in individuals using the intervention versus the control toothpaste for 6 months.
Blood Pressure Change | 6 months
  Does blood pressure change at all in individuals using the intervention versus the control toothpaste for 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Zoe Brookes, BDS, MJDF, PCHE, SFHEA, PhD, Principal Investigator — University of Plymouth
Locations (1):
- Derriford Dental Education Facility, Plymouth, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All outcome measures will be published however, there will be no way of linking data back to individual patients.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: These will all be made available at the end of the study through publication, as the University of Plymouth own the independent data produced via this collaborative project.
Access Criteria: Online access unrestricted